CLINICAL TRIAL: NCT02141919
Title: A Phase II Trial of Stereotactic Ablative Body Radiation Therapy (SABR) for Patients With Primary Renal Cancer (RCC)
Brief Title: Stereotactic Ablative Body Radiation Therapy for Patients With Primary Renal Cancer
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Principal Investigator, Raquibul Hannan, Associate Professor of Medicine, University of Texas Southwestern Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STU 122013-030
Record Dates: First submitted 2014-05-12; First posted 2014-05-20 (Estimated); Last update posted 2025-12-26 (Actual); Status verified 2025-12

CONDITIONS: Renal Cancers
Keywords: renal cancer
MeSH Terms: conditions — Kidney Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Stereotactic Ablative Radiation Therapy (Experimental): Stereotactic Ablative Radiation Therapy (SABR)
  Interventions: Radiation: Stereotactic Ablative Radiation Therapy

INTERVENTIONS:
Radiation: Stereotactic Ablative Radiation Therapy — Stereotactic Ablative Body Radiation Therapy (SABR): 3 fractions of 12Gy, or 4 fractions of 10Gy or 5 fractions of 8 Gy
  Other Names: SABR

SUMMARY:
The goal of this phase II clinical trial is to evaluate the efficacy of the completely non-invasive treatment option of stereotactic radiation therapy for the treatment of biopsy proven and growing small renal tumors.

DETAILED DESCRIPTION:
Current treatment options for primary renal cancer include surgery or ablative techniques-all are invasive or minimally invasive options. The completely noninvasive treatment option of stereotactic radiation therapy (SABR), which has become standard of care in many cancer sites, has not been explored for primary renal cancer. With multiple technological advances, it is now feasible to safely treat a moving intra-abdominal tumor such as that in a kidney. This proposed clinical trial evaluates the efficacy of SABR in treating patients with early renal cancers. Growing renal masses will first be biopsied to confirm the diagnosis of renal cancer. Patients will then undergo treatment with SABR of 3-5 fractions completing within three weeks. Treatment response will be evaluated using sequential MRI scans and a second tumor biopsy one year after treatment. Monitoring of treatment toxicity and kidney function will also be performed.

ELIGIBILITY:
Inclusion Criteria

* Age ≥ 18 years.
* Renal mass ≤ 5cm

  * The treating renal mass must be ≤ 5cm. Other renal masses (cysts etc.) of any size will not make the subject ineligible
* Biopsy proven Renal neoplasm

  * All histology of renal cancers are included including oncocytoma
* Growth of renal mass >2mm in radiographic scans must be demonstrated within a one year period.
* Ability to understand and the willingness to sign a written informed consent.
* Subject is able to undergo either an MRI or administration of contrast agent for CT
* Women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) for the duration of the study. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately.
* A female of child-bearing potential is any woman (regardless of sexual orientation, having undergone a tubal ligation, or remaining celibate by choice) who meets the following criteria:

  * Has not undergone a hysterectomy or bilateral oophorectomy; or
  * Has not been naturally postmenopausal for at least 12 consecutive months (i.e., has had menses at any time in the preceding 12 consecutive months).

Exclusion Criteria:

* Subject has received any treatment for the treating renal mass; such as RFA or cyroablation.

  * If other renal masses received RFA or cryoablation or surgery, then these patients are eligible.
* Subjects received previous abdominal radiation
* Evidence of Metastatic Disease, unless disease-free for ≥ 3 years prior to registration, (non-melanomatous skin cancer and in-situ cancers are okay).
* Female subjects who are pregnant or planning to become pregnant during the course of SABR.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2013-06 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Eliminate its growth and tumor viability. | 2 years
  To evaluate if SABR to small renal tumors is able to eliminate its growth and viable tumor.

SECONDARY OUTCOMES:
Adverse events | 2 years
  To describe the adverse events associated with the administration of SABR to renal tumors.
growth rate of renal tumors | 2 years
  To measure the growth rate of renal tumors after SABR treatment.
Renal function | 2 years
  To measure the changes in kidney function, creatinine levels, renal perfusion and GFR after SABR treatment
Tumor Viability | one year
  To measure tumor viability pathologically one year after SABR treatment with biopsy.
progression of disease | 2 years
  To assess radiographic changes to the renal tumor after SABR treatment including tumor viability, enhancement necrosis,T2 tumor cellularity with diffusion-weighted imaging. To assess local, regional and systemic progression of disease after SABR to SRM .To assess time to progression (TTP) of disease from the first SABR treatment.
  To assess progression free survival (PFS). PFS is defined as the length of time from start of treatment to the time of loco-regional disease progression or death from any cause.
  To assess overall survival (OS). OS is defined as the duration of time from start of treatment to the time of death from any cause.
  To assess tumor growth, local failure and indeterminate disease response (IDR).

CONTACTS AND LOCATIONS:
Overall Officials: Raquibul Hannan, MD, PhD, Principal Investigator — UTSW
Locations (1):
- University of Texas Southwestern, Dallas, Texas, United States

DOCUMENTS (1):
  • Study Protocol (2020-05-19): https://cdn.clinicaltrials.gov/large-docs/19/NCT02141919/Prot_000.pdf